CLINICAL TRIAL: NCT05004532
Title: Efficacy of Preoperative Transversus Abdominis Plane Block in Acute Appendicitis Pain and Its Success in Postoperative Pain
Brief Title: Transversus Abdominis Plane Block in Acute Appendicitis Pain Managment
Status: Completed | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, HULYA TOPCU, assistant professor M.D. Hulya TOPCU, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 19/08/2020 - 223
Record Dates: First submitted 2021-06-04; First posted 2021-08-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Acute Appendicitis; Acute Abdomen; Postoperative Pain
Keywords: transversus abdominis plane nerve block; acute appendicitis; acute pain; postoperative pain
MeSH Terms: conditions — Appendicitis; Abdomen, Acute; Pain, Postoperative; Acute Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, it was aimed to investigate the analgesic efficacy of the preoperatively applied Transversus Abdominis Plane (TAP) Block in the management of acute appendicitis-related abdominal pain and post-appendectomy pain.

DETAILED DESCRIPTION:
TAP block creates an analgesic effect by blocking both sensory skin dermotams and viscerosomatic transmission. TAP block with ultrasound was first performed by Hebbard, and the use of USG made the procedure faster and safer. TAP block has been successfully applied for analgesia in procedures such as laparoscopic colocystectomy, inguinal hernia repair, abdominal hysterectomy, prostatectomy and appendectomy. According to the surgical incision to be applied, TAP block is performed from different anatomical regions. It is also applied for pain palliation in intra-abdominal etiologies or rarely for anesthesia in surgical procedures.

The analgesic efficacy of TAP block on preoperative abdominal pain and postoperative surgical pain in acute appendicitis was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with a diagnosis of acute appendicitis,
* with abdominal pain,
* tap block applied for perioperative pain management.

Exclusion Criteria:

* The data of patients who underwent laparoscopic appendectomy
* additional surgical procedure other than appendectomy (right hemicolectomy, etc.)
* who were diagnosed other than acute appendicitis after the surgical procedure (diverticulitis, tumor, etc.),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who underwent open appendectomy with the diagnosis of acute appendicitis, who underwent TAP block, were identified retrospectively. Demographic data of the patients, change of pain scores at rest and with coughing, postoperative pain scores, postoperative analgesic need were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Verbal Numerical Pain Scale | postoperative time 24 hour time
  <4 good pain managment , >4-10 bad pain managment

SECONDARY OUTCOMES:
BMI | preoperative
  kg/(m2)
weight | preoperative
  kg

IPD SHARING:
Plan to Share IPD: No